CLINICAL TRIAL: NCT03576924
Title: The Power of Choice on Autonomy Support, Motivation, Exercise Adherence and Cardiorespiratory Fitness Among Adults With Elevated Blood Glucose
Brief Title: Power of Choice on Autonomy, Motivation, Exercise Adherence, and Cardiorespiratory Fitness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Mary Jung, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: G-18-0022225
Record Dates: First submitted 2018-06-21; First posted 2018-07-05 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Elevated Blood Sugar
Keywords: Autonomy Support; Exercise Motivation; Physical Activity Adherence; Cardiorespiratory Fitness; Prediabetes
MeSH Terms: conditions — Hyperglycemia; Prediabetic State

STUDY DESIGN:
Intervention Model Description: This is a single-centre, 3-arm parallel-group randomized trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MICT (Active Comparator): Continuous exercise for 30 minutes per session at 60-70% of heart rate max for five times per week, consistent with physical activity guidelines that advocate 150 minutes per week of moderate activity.
  Interventions: Behavioral: MICT
- HIIT (Active Comparator): Five repeated vigorous intervals of 1-min duration at 80-90% of heart rate max interspersed with 1-min recovery periods; 3-min warm-up and 2-min cool-down, making the total session duration 15 minutes for five times/week, equated to match the guidelines of 75 min of vigorous exercise per week.
  Interventions: Behavioral: HIIT
- CHOICE (Experimental): Participants will be introduced to HIIT and MICT during sessions 1 and 2 of the 4-week intervention in a counterbalanced randomized order, and will thereafter self-select one of the two exercise types for remaining sessions. Exercise will be matched to the parallel imposed conditions.
  Interventions: Behavioral: CHOICE

INTERVENTIONS:
Behavioral: MICT — Individuals randomized to MICT will be asked to engage in only MICT 5 times/week for 30 min/session at 60-70% of heart rate max, consistent with physical activity guidelines of 150 min/week of moderate activity. Individuals are asked to engage in only MICT exercise during the 4-week supervised and unsupervised exercise sessions. During the supervised exercise the intensity will be based on the heart rate (HR) monitors and psychophysiological responses of perceived exertion. The exercise training is paired with 30-50 minutes of behavioral counselling that is identical for all three interventions.
  Arms: MICT
Behavioral: HIIT — Individuals randomized to HIIT will be asked to engage in only HIIT 5 times/week for 4 weeks. HIIT consists of 5 repeated vigorous intervals of 1-min duration at 80-90% of heart rate max interspersed with 1-min recovery periods. A 3-min warm-up and 2-min cool-down are also included, for a total session duration of 15 minutes. This matches the guidelines of 75 min of vigorous exercise per week. During the supervised exercise sessions, intensity will be based on HR monitors and psychophysiological responses of perceived exertion. The exercise training is paired with 30-50 minutes of behavioral counselling that is identical for all three interventions.
  Arms: HIIT
Behavioral: CHOICE — Participants will first be familiarized with HIIT and MICT in a randomized, counter-balanced order during supervised sessions 1 and 2, and will subsequently self-select the exercise type for the supervised and unsupervised exercise sessions. The HIIT and MICT protocols will match to the parallel imposed conditions. During the supervised exercise, intensity will also be based on HR monitors and psychophysiological responses of perceived exertion. The exercise training is paired with 30-50 minutes of behavioral counselling that is identical for all three interventions.
  Arms: CHOICE

SUMMARY:
People with elevated blood sugar levels are at increased risk of developing chronic medical conditions such as obesity, type 2 diabetes, and cardiovascular disease. Improving cardiorespiratory fitness (CRF) in adults with elevated blood sugar levels is important for preventing the onset of such medical conditions. The primary aim of this study is to determine whether providing a choice between two different types of exercise in a diabetes prevention intervention improves perceived autonomy, exercise motivation, physical activity behavior, and subsequently CRF to a greater extent than imposed exercise among adults with elevated blood sugar.

DETAILED DESCRIPTION:
This trial has been informed by self-determination theory. The theory states that individuals who choose their own activities report increased autonomy and internal reasons/motivations to change a behavior as opposed to external reasons (to satisfy another person's suggestions). Perceived autonomy support and internal motivation for performing a behavior are linked with improved long-term adherence to the behavior change, which subsequently leads to physiological adaptations such as an increase in CRF.

The primary outcome of this study is participants' perceived autonomy support after a 4-week diabetes prevention program. The secondary outcomes are 1) changes in exercise-related motivation from baseline to immediately post-intervention and 6-months post-intervention, 2) physical activity behavior 6-months post-intervention while controlling for baseline values, and 3) CRF 6-months post-intervention while controlling for baseline values. Seventy-seven low-active adults between 18-75 years of age with elevated blood sugar levels (HbA1c between 5.7%-6.4% or American Diabetes Association risk assessment >5) have been randomized to a 4-week supervised intervention involving behavioral counseling and one of three exercise conditions: 1) imposed high-intensity interval training (HIIT; n=26); 2) imposed moderate-intensity continuous training (MICT; n=26), or 3) choice between MICT or HIIT (CHOICE; n=24). It is hypothesized that when compared to HIIT and MICT, the CHOICE condition will have greater perceived autonomy support immediately after the 4-week intervention, display more internal motivation immediately after the 4-week intervention, and show greater improvements in physical activity adherence and CRF 6-months post-intervention. This proposed trial will provide theory- and evidence-based information whether providing choice for engaging in HIIT or MICT is associated with greater improvements in perceived autonomy support, motivation regulation, physical activity behavior, and CRF.

ELIGIBILITY:
Inclusion Criteria:

* BMI 22-45 kg/m2;
* HbA1c score indicative of elevated blood sugar (5.7-6.4%);
* Blood pressure of <160/99 mm Hg assessed according to Canadian Hypertension Education Program guidelines;
* Without diagnosed diabetes;
* No prior history of cardiovascular disease;
* Not on hormone replacement therapy;
* Not on beta-blockers;
* Cardiovascular medications (e.g., statins) will be allowed if patients are on stable therapy (6 months on same dose)

Exclusion Criteria:

* Taking glucose-lowering medications (i.e. metformin);
* Any explicit contraindications to exercise (e.g., musculoskeletal injury)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E. Jung, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Little JP, Safdar A, Wilkin GP, Tarnopolsky MA, Gibala MJ. A practical model of low-volume high-intensity interval training induces mitochondrial biogenesis in human skeletal muscle: potential mechanisms. J Physiol. 2010 Mar 15;588(Pt 6):1011-22. doi: 10.1113/jphysiol.2009.181743. Epub 2010 Jan 25. PMID 20100740
- [Background] Little JP, Gillen JB, Percival ME, Safdar A, Tarnopolsky MA, Punthakee Z, Jung ME, Gibala MJ. Low-volume high-intensity interval training reduces hyperglycemia and increases muscle mitochondrial capacity in patients with type 2 diabetes. J Appl Physiol (1985). 2011 Dec;111(6):1554-60. doi: 10.1152/japplphysiol.00921.2011. Epub 2011 Aug 25. PMID 21868679
- [Background] Hood MS, Little JP, Tarnopolsky MA, Myslik F, Gibala MJ. Low-volume interval training improves muscle oxidative capacity in sedentary adults. Med Sci Sports Exerc. 2011 Oct;43(10):1849-56. doi: 10.1249/MSS.0b013e3182199834. PMID 21448086
- [Background] Kodama S, Saito K, Tanaka S, Maki M, Yachi Y, Asumi M, Sugawara A, Totsuka K, Shimano H, Ohashi Y, Yamada N, Sone H. Cardiorespiratory fitness as a quantitative predictor of all-cause mortality and cardiovascular events in healthy men and women: a meta-analysis. JAMA. 2009 May 20;301(19):2024-35. doi: 10.1001/jama.2009.681. PMID 19454641
- [Background] O'Donovan G, Owen A, Bird SR, Kearney EM, Nevill AM, Jones DW, Woolf-May K. Changes in cardiorespiratory fitness and coronary heart disease risk factors following 24 wk of moderate- or high-intensity exercise of equal energy cost. J Appl Physiol (1985). 2005 May;98(5):1619-25. doi: 10.1152/japplphysiol.01310.2004. Epub 2005 Jan 7. PMID 15640382
- [Background] Jung ME, Bourne JE, Little JP. Where does HIT fit? An examination of the affective response to high-intensity intervals in comparison to continuous moderate- and continuous vigorous-intensity exercise in the exercise intensity-affect continuum. PLoS One. 2014 Dec 8;9(12):e114541. doi: 10.1371/journal.pone.0114541. eCollection 2014. PMID 25486273
- [Background] Jung ME, Bourne JE, Beauchamp MR, Robinson E, Little JP. High-intensity interval training as an efficacious alternative to moderate-intensity continuous training for adults with prediabetes. J Diabetes Res. 2015;2015:191595. doi: 10.1155/2015/191595. Epub 2015 Mar 30. PMID 25918728
- [Background] National Research Council (US) Panel on Handling Missing Data in Clinical Trials. The Prevention and Treatment of Missing Data in Clinical Trials. Washington (DC): National Academies Press (US); 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK209904/ PMID 24983040
- [Background] Preacher KJ, Hayes AF. SPSS and SAS procedures for estimating indirect effects in simple mediation models. Behav Res Methods Instrum Comput. 2004 Nov;36(4):717-31. doi: 10.3758/bf03206553. PMID 15641418

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MICT | HIIT | CHOICE
Started | 26 | 27 | 24
Completed | 24 | 24 | 21
Not Completed | 2 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MICT | HIIT | CHOICE | Total
Number analyzed (Participants) | 26 | 27 | 24 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (11.9) | 62.4 (9.2) | 62.3 (7.8) | 61.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 19 | 58
  Male | 7 | 7 | 5 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 26 | 27 | 24 | 77

OUTCOME MEASURES:

1. Primary Outcome: Perceived Autonomy Support
Description: Individual participants' perceived autonomy support will be measured using the Learning Climate Questionnaire (LCQ) adapted by Williams and Deci. The LCQ is a 15-item self-report questionnaire that measures perceived autonomy support and has been previously validated and shown to have strong internal reliability. The questionnaire uses a 7-point Likert scale ranging from 1 "strongly disagree" to 7 "strongly agree". For this study, the anchoring questions are modified to replace the term "instructor" with "coach". Scoring of individual results is done by averaging individual responses after reverse-coding item #13, with a minimum score of 1 and a maximum score of 7. Higher scores indicate a higher perception of autonomy support.
Time Frame: Four weeks post-intervention.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | MICT | HIIT | CHOICE
Number analyzed (Participants) | 24 | 24 | 21
score on a scale | 6.78 [6.32 to 7] | 6.85 [6.30 to 7] | 6.77 [6.21 to 7]

2. Secondary Outcome: Change in Exercise Motivation Regulation
Description: Participants' change in motivation regulation from baseline to post-intervention and subsequently 6 months later is measured using the Behavioral Regulation in Exercise Questionnaire-2 (BREQ-2). The BREQ-2 is a 19-item self-report questionnaire that measures one's motivation to exercise. The questionnaire uses a 5-point Likert scale ranging from 0 "not true for me" to 4 "very true for me". The relative autonomy index (RAI) is used to provide an index of the degree to which participants feel self-determined ranging from a minimum score of -24 to a maximum score of +20, with higher positive scores indicating more autonomous forms of motivation regulation. The RAI is calculated by first averaging each subscale, then multiplying each average by a subscale weighting, and subsequently summing the weighted subscale scores. Weighting for each subscale are as follows: amotivation (-3), external regulation (-2), introjected regulation (-1), identified regulation (+2), intrinsic regulation (+3).
Time Frame: Baseline, four weeks post-intervention, and 6 months post-intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | MICT | HIIT | CHOICE
Number analyzed (Participants) | 24 | 24 | 21
score on a scale
  Baseline | 10.0 [7.1 to 12.9] | 10.1 [6.7 to 13.6] | 8.9 [5.4 to 12.4]
  Post-Intervention | 11.7 [8.8 to 14.7] | 11.4 [8.0 to 14.8] | 10.8 [7.2 to 14.4]
  6-Month Follow-Up | 11.1 [7.7 to 14.4] | 10.7 [7.3 to 14.1] | 10.6 [7.0 to 14.2]

3. Secondary Outcome: Change in Physical Activity Behavior (Self-Report)
Description: Change in physical activity behavior from baseline to 6 months later will be measured using the Godin Leisure-Time Exercise Questionnaire (GLTEQ). The GLTEQ requires individuals to report their frequency of engaging in strenuous, moderate, and mild exercise during a typical week in bouts of 15 minutes or longer. Scoring of the GLTEQ consists of first multiplying reported frequencies by their related metabolic equivalent (MET) values (strenuous: 9METs, moderate: 5METs, mild: 3METs), and then summing the products for a total score. Interpretation of the scores follows the categories proposed by Godin, where a score of 24 units or higher indicates an individual is active, a score between 14 and 23 indicates an individual is moderately active, and a score below 14 indicates an individual is insufficiently active. The minimum score is 0 and there is no maximum score. Higher scores indicate higher levels of physical activity behavior.
Time Frame: Baseline, 6-months after the intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | MICT | HIIT | CHOICE
Number analyzed (Participants) | 24 | 24 | 21
score on a scale
  Baseline | 21.2 [8.4 to 33.9] | 27.5 [12.2 to 42.9] | 27.8 [12.7 to 42.9]
  6-Month Follow-Up | 37.1 [22.4 to 51.8] | 35.0 [20.4 to 49.7] | 44.6 [28.9 to 60.4]

4. Secondary Outcome: Change in Physical Activity Behavior (Accelerometry)
Description: Change in physical activity behavior from baseline to 6 months later will also be measured using 7-day triaxial accelerometry data. Participants wear an Actigraph GT3X-BT for seven consecutive days at the top of their right hip at a sampling rate of 100Hz. Accelerometry data is considered valid if the participant wears the accelerometer for a minimum of 10 hours/day and at least 4 of the 7 days of the week. Non-wear time is defined as any period of 60 minutes or longer with no recorded activity counts. Physical activity is measured by summing activity counts in 60-second epochs, and cut-off activity count thresholds for defining intensity follows Troiano and colleagues' convention. Free-living physical activity behavior is operationalized as average daily minutes of MVPA and is calculated by summing both moderate and vigorous activity count minutes and subsequently dividing by the number of valid wear days.
Time Frame: Baseline, 6 months after the intervention
Measure: Mean (95% Confidence Interval); unit: minutes/day
Arm/Group | MICT | HIIT | CHOICE
Number analyzed (Participants) | 24 | 24 | 21
minutes/day
  Baseline | 31.9 [15.3 to 48.6] | 40.5 [24.6 to 56.3] | 38.9 [21.1 to 56.7]
  6-Month Follow-Up | 29.5 [12.7 to 46.3] | 32.9 [16.4 to 49.4] | 34.5 [16.7 to 52.4]

5. Secondary Outcome: Change in Physical Activity Behavior (Fitbit)
Description: A wearable activity tracker (Fitbit Luxe™) is also provided to each participant to track change in physical activity behavior from baseline to 6 months later in free-living conditions. We define a valid wear day as any day with a minimum of 10 hours of wear time determined by continuous minute-by-minute heart rate recordings. Non-wear time is defined as a period of 60 continuous minutes with no heart rate recordings. A minimum of 4 out of 7 consecutive days of the week are required for the week to be considered valid. Free-living physical activity behavior is operationalized as average daily minutes of MVPA and is calculated by summing the daily minutes spent in moderate and intense activities per day and subsequently dividing by the number of valid wear days. Activity intensity levels are determined by using Fitbit-derived algorithms, and number of minutes per day at each intensity level are imported into Fitabase.
Time Frame: Baseline, 6 months after intervention
Measure: Mean (95% Confidence Interval); unit: minutes/day
Arm/Group | MICT | HIIT | CHOICE
Number analyzed (Participants) | 24 | 24 | 21
minutes/day
  Baseline | 71.4 [47.6 to 95.2] | 70.4 [47.8 to 93.1] | 68.7 [43.2 to 94.2]
  6-Month Follow-Up | 63.7 [38.9 to 88.6] | 61.8 [37.1 to 86.5] | 56.9 [31.6 to 82.2]

6. Secondary Outcome: Change in Cardiorespiratory Fitness
Description: Participants' change in cardiorespiratory fitness (CRF) from baseline to 6 months later is calculated based on the minutes and seconds participants are able to achieve in submaximal 12-lead ECG stress tests performed at a cardiac rehabilitation clinic. Calculation of CRF is conducted according to Bruce and colleagues' equation for estimated maximal volume of oxygen intake (VO2max) in mL/(kg*min). Calculations are stratified by biological sex, where w is the weighting factor for sex (1=men; 2=women) and t is the duration of the protocol in seconds:
  VO2max=6.70-2.82w+0.056t
Time Frame: Baseline, 6 months after intervention
Measure: Mean (95% Confidence Interval); unit: mL/min/kg
Arm/Group | MICT | HIIT | CHOICE
Number analyzed (Participants) | 24 | 24 | 21
mL/min/kg
  Baseline | 35.4 [29.2 to 41.5] | 35.4 [29.5 to 41.4] | 35.9 [29.3 to 42.5]
  6-Month Follow-Up | 38.1 [31.9 to 44.2] | 36.7 [30.7 to 42.7] | 38.0 [31.4 to 44.6]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | MICT | HIIT | CHOICE
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27 | 0/24
Other Adverse Events (participants affected / at risk) | 0/26 | 2/27 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MICT (N=26) | HIIT (N=27) | CHOICE (N=24)
Back Surgery (Surgical and medical procedures) | 0 | 1 | 0 — Back surgery was unrelated to the current study.
Cancer (General disorders) | 0 | 1 | 0 — Diagnosis was not related to the current study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-03): https://cdn.clinicaltrials.gov/large-docs/24/NCT03576924/Prot_SAP_000.pdf